CLINICAL TRIAL: NCT06129487
Title: Evaluations of Alcohol Warning Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Oakland University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zexin Ma, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2023-0021; 7R03CA273391-02 (NIH)
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Oral Cancer; Esophageal Cancer; Larynx Cancer; Alcohol Drinking
MeSH Terms: conditions — Mouth Neoplasms; Esophageal Neoplasms; Laryngeal Neoplasms; Alcohol Drinking | interventions — Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Pictorial Warning Labels (Experimental): Participants in this arm will be presented with three narrative pictorial warning labels for alcoholic beverages.
  Interventions: Behavioral: Narrative pictorial warning labels for alcoholic beverages
- Non-Narrative Pictorial Warning Labels (Experimental): Participants in this arm will be presented with three non-narrative pictorial warning labels for alcoholic beverages.
  Interventions: Behavioral: Non-narrative pictorial warning labels for alcoholic beverages

INTERVENTIONS:
Behavioral: Narrative pictorial warning labels for alcoholic beverages — Pictorial warning labels consisting of text and narrative imagery (e.g., photos of cancer patients) conveying the risk of alcohol for oral cancer, esophageal cancer, and larynx cancer.
  Arms: Narrative Pictorial Warning Labels
Behavioral: Non-narrative pictorial warning labels for alcoholic beverages — Pictorial warning labels consisting of text and non-narrative imagery (e.g., images of diseased organs) conveying the risk of alcohol for oral cancer, esophageal cancer, and larynx cancer.
  Arms: Non-Narrative Pictorial Warning Labels

SUMMARY:
The goal of this study is to determine the effectiveness of pictorial warning labels (PWLs) featuring narrative (vs. non-narrative) content in communicating the cancer risk of alcohol. Participants will be randomized to view either three narrative or non-narrative PWLs. Key outcome variables include visual attention, message reactance, risk perceptions, and intentions to reduce and stop drinking.

DETAILED DESCRIPTION:
The goal of this study is to determine the effectiveness of pictorial warning labels (PWLs) featuring narrative (vs. non-narrative) content in communicating the cancer risk of alcohol. Participants will be recruited from online panels. Participants will first be invited to participate in an online screening survey. Eligible participants will be invited to participate in the main experiment. In the main experiment, participants will first answer questions concerning baseline alcohol consumption and other background information. Then they will engage with a webcam-based eye-tracking task through Sticky by Tobii. Participants will first read instructions and tips related to completing the eye-tracking task. They will complete a brief calibration procedure and be presented with either three narrative PWLs or three non-narrative PWLs. Sticky by Tobii will record participants' gaze, thereby measuring visual attention to each PWL. After viewing each PWL, participants will answer a few questions. After viewing all three PWLs, they will answer questions based on all images combined. Upon study completion, participants will be compensated. A follow-up survey will be sent to participants after two weeks, which includes questions about their drinking behaviors, information seeking behaviors, and social interactions.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 21 years old;
2. have consumed more than three alcoholic drinks per week over the past year;
3. be willing to participate in remote eye tracking tasks and have necessary technical support to complete remote eye tracking tasks (i.e., having access to high-speed Internet and a computer/tablet/phone equipped with a high-speed camera).

Exclusion Criteria:

1. be younger than 21 years old;
2. has not consumed more than three alcoholic drinks per week over the past year;
3. be not willing to participate in remote eye tracking tasks and have no necessary technical support to complete remote eye tracking tasks (i.e., having access to high-speed Internet and a computer/tablet/phone equipped with a high-speed camera).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zexin Ma, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- Online Survey-Experiment, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified dataset, study protocol, sample informed consent, and data dictionary will be made available to the research community free of charge through ICPSR (https://www.openicpsr.org/).
Supporting Information: Study Protocol, ICF
Time Frame: Datasets will be shared upon the publication of the manuscripts and will be available to the research community in perpetuity.
Access Criteria: All de-identified study data use will be made available as public use data to the research community through ICPSR. Users of the public use data must register with ICPSR and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.

RESULTS

PARTICIPANT FLOW:
Groups:
- Narrative Pictorial Warning Labels: Participants in this arm were presented with three narrative pictorial warning labels (PWLs) for alcoholic beverages. Narrative PWLs included a photo showing the lived experiences of individuals affected by alcohol-related cancer (e.g., a headshot of a man with a misshapen jaw) and a text warning statement (e.g., WARNING: Drinking alcohol can cause oral cancer). The warnings focused on oral, esophageal, and laryngeal cancers, respectively.
- Non-Narrative Pictorial Warning Labels: Participants in this arm will be presented with three non-narrative pictorial warning labels (PWLs) for alcoholic beverages. Non-narrative PWLs contained graphic images of diseased organs (e.g., a closeup image of a mouth with rotten teeth and oral thrush) and a text warning statement (e.g., WARNING: Drinking alcohol can cause oral cancer). The warnings focused on oral, esophageal, and laryngeal cancers, respectively.
Period: Overall Study
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Started | 526 | 527
Completed | 328 | 321
Not Completed | 198 | 206
Not completed — Data loss was due to technical issues related to eye tracking. | 198 | 206

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels | Total
Number analyzed (Participants) | 328 | 321 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.68 (11.66) | 40.41 (12.15) | 39.54 (11.93)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at birth: Female | 152 | 131 | 283
  Sex at birth: Male | 174 | 188 | 362
  Sex at birth: Prefer not to say | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 42 | 83
  Not Hispanic or Latino | 287 | 279 | 566
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 18 | 17 | 35
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 39 | 44 | 83
  White | 251 | 238 | 489
  More than one race | 16 | 20 | 36
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dwell Time
Description: Dwell time measures the total duration of attention to an area of interest (AOI). Each warning label consisted of two AOIs: image AOI and text AOI. Dwell time for each AOI was averaged across three PWLs within each arm.
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Population: Sticky's internal algorithms determined cases where the eye tracking data is less than "perfect" and only returns "usable" data. Thus, only usable eye tracking data were analyzed.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 192 | 213
seconds | 8.75 (0.069) | 8.47 (0.066)

2. Primary Outcome: Visit Count
Description: Visit count measures the total number of times participants viewed an area of interest (AOI). Each warning label consisted of two AOIs: image AOI and text AOI. Visit count for each AOI was averaged across three PWLs within each arm.
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: visit
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 192 | 213
visit | 13.74 (0.443) | 13.58 (0.420)

3. Primary Outcome: Reactance
Description: Reactance were measured after exposure to each PWL (i.e., three times in total). It was assessed using the brief Reactance to Health Warnings Scale (Hall et al., 2017). Participants were asked to indicate how much each warning tried to manipulate them, annoyed them, and was overblown (1 = not at all, 5 = a great deal). Reactance for each PWL was averaged across three PWLs within each arm.
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 327 | 318
score on a scale | 2.38 (0.055) | 2.54 (0.055)

4. Primary Outcome: Affective Risk Perceptions
Description: Affective risk perceptions were assessed once after participants viewed all three PWLs. Participants were asked to indicate how worried they are about getting a specific type of cancer if they keep drinking the amount of alcohol like they do now. Participants responded on a five-point scale (1 = Not at all worried, 2=Slightly worried, 3=Moderately worried, 4=Very worried, 5=Extremely worried).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 2.27 (0.062) | 2.38 (0.063)

5. Primary Outcome: Experiential Risk Perceptions
Description: Experiential risk perceptions were assessed once after participants viewed all three PWLs. Participants were asked to indicate how vulnerable they feel about getting a specific type of cancer if they keep drinking the amount of alcohol like they do now. Participants responded on a five-point scale (1 = Not at all vulnerable, 2=Slightly vulnerable, 3=Moderately vulnerable, 4=Very vulnerable, 5=Extremely vulnerable).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 2.35 (0.058) | 2.46 (0.058)

6. Primary Outcome: Perceived Susceptibility
Description: Perceived susceptibility were assessed once after participants viewed all three PWLs. Participants were asked to indicate how likely it is that they will get a specific type of cancer if they keep drinking the amount of alcohol like they do now. Participants responded on a five-point scale (1 = Not at all likely, 2=A little likely, 3=Somewhat likely, 4=Very likely, 5=Extremely likely).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 2.072 (0.053) | 2.102 (0.054)

7. Primary Outcome: Comparative Risk
Description: Comparative risk were assessed once after participants viewed all three PWLs. Participants were asked to indicate compared to an average person their age, race, and sex, how likely do they think they will get a specific type of cancer if they keep drinking the amount of alcohol like they do now. Participants responded on a five-point scale (1=Much less likely, 2=Less likely, 3=About as likely, 4=More likely, 5=Much more likely).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 2.71 (0.056) | 2.85 (0.057)

8. Primary Outcome: Perceived Severity of Harm
Description: Perceived severity of harm were assessed once after participants viewed all three PWLs. Participants were asked to indicate how much getting a specific type of cancer because of drinking would affect their life. Participants responded on a five-point scale (1=Not at all, 2=Very little, 3=Somewhat, 4=Quite a bit, 5=A great deal).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 4.47 (0.05) | 4.55 (0.05)

9. Primary Outcome: Intentions to Reduce Drinking
Description: Intentions to reduce drinking were assessed once after participants viewed all three PWLs. Participants were asked to answer questions such as "How interested are you in reducing drinking in the next 6 months?" Participants responded to these questions on an appropriately labeled 5-point scale (e.g., 1 = Not at all interested, 2=Slightly interested, 3=Moderately interested, 4=Very interested, 5=Extremely interested).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 3.08 (0.05) | 3.14 (0.05)

10. Primary Outcome: Intentions to Stop Drinking
Description: Intentions to stop drinking were assessed once after participants viewed all three PWLs. Participants were asked to answer three questions such as "How interested are you in stopping drinking in the next 6 months?" Participants responded to these questions on an appropriately labeled 5-point scale (e.g., 1 = Not at all interested, 2=Slightly interested, 3=Moderately interested, 4=Very interested, 5=Extremely interested).
Time Frame: Assessed during the one-time 15-minute online survey experiment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
Number analyzed (Participants) | 328 | 321
score on a scale | 2.26 (0.068) | 2.37 (0.069)
Statistical Analysis 1: Comparison: Narrative Pictorial Warning Labels vs Non-Narrative Pictorial Warning Labels; Test type: Superiority; p = 0.256, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed for this online survey experiment.
Description: Deaths and/or adverse events were not monitored/assessed as this was an online study where participants completed the survey on their own computer at a location of their choice.
Arm/Group | Narrative Pictorial Warning Labels | Non-Narrative Pictorial Warning Labels
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT06129487/Prot_SAP_000.pdf